CLINICAL TRIAL: NCT02016521
Title: "Keep Cool": a Randomized Trial on the Effect of Wearing a Garment Made of Cooling Fabrics on Thermoregulatory, Cardiorespiratory, and Perceptual Responses to Exercise in Endurance-trained Athletes
Brief Title: Cooling Fabrics and Exercise Performance in Endurance Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Assistant Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A00-M108-13A
Record Dates: First submitted 2013-12-15; First posted 2013-12-20 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Cooling Fabrics; Exercise Performance; Thermoregulation
Keywords: Exercise; Clothing; Core body temperature; Skin Temperature; Performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cooling Fabric (Experimental): Garment made of 100% nylon fabric consisting of long sleeved shirt and full trouser.
  Interventions: Other: Cooling Fabric
- Placebo Garment (Placebo Comparator): Garment made of 100% polyester consisting of long sleeved shirt and full trouser.
  Interventions: Other: Placebo Garment

INTERVENTIONS:
Other: Cooling Fabric — Garment made of 100% nylon and consisting of long sleeved shirt and full trouser.
  Arms: Cooling Fabric
Other: Placebo Garment — Garment made of 100% polyester consisting of long sleeved shirt and full trouser
  Arms: Placebo Garment

SUMMARY:
In humans, the primary means of cooling the body during exercise is through the evaporation of sweat from the skin surface. Clothing represents a layer of insulation that hinders the evaporation of sweat from the surface of the skin. It follows that clothing that imposes the least amount of resistance to evaporative heat loss may prove beneficial to the thermoregulatory, physiological and perceptual response to exercise, particularly in elite endurance-trained athletes. Thus, the purpose on this study is to examine the influence of wearing a sportswear garment made of a fabric (100% nylon) with superior evaporative characteristics on detailed thermoregulatory, cardiorespiratory, metabolic and perceptual responses to maximal exercise testing at normal room temperature and relatively humidity in a group of 25 endurance-trained cyclists and triathletes aged 20-60 years. It is hypothesized that wearing a garment made of 100% nylon will improve exercise performance (e.g., exercise endurance time) and that this improvement will reflect improvements in thermoregulatory, cardiorespiratory, metabolic and perceptual responses to exercise. Athletes will be recruited via contact with coaches of the McGill University Cycling and Triathlon teams as well as through contact with coaches of competitive cycling and triathlon teams/training groups in the Montreal and surrounding area. Initial contact will consist of a thorough explanation of the study procedures and pre-screening for the inclusion/exclusion criteria prior to study consent by the Principal Investigator and/or his delegate, either in person or by telephone or email. Eligible participants will visit McGill's Clinical Exercise & Respiratory Physiology Laboratory on 3 separate occasions over a period of 10-14 days. Visit 1 will include a maximal incremental bicycle exercise test for familiarization purposes and to determine maximal power output (MPO). Visits 2 and 3 will include a constant-power-output bicycle exercise test at 85% MPO under one of two conditions, in randomized order: (1) while wearing a garment made of 100% polyester, i.e., placebo; and (2) while wearing a garment made of 100% nylon, i.e., cooling fabric. At rest and during exercise at visits 2 and 3, detailed assessments of core body temperature will be made using a temperature sensor placed into the esophagus, while skin temperature and other physiological and perceptual parameters will be measured using standard techniques.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Non-smoker
* Aged 20-60 years
* Competitive cyclist and/or triathlete competing at the regional, provincial, national and/or international level.
* Maximal rate of oxygen uptake on incremental cycle exercise testing greater than or equal to 60 ml/kg/min.
* Forced expiratory volume in 1 second greater than or equal to 80% predicted.
* Forced expiratory volume in 1 second/forced vital capacity ratio greater than or equal to 70%.
* Women: taking an oral contraceptive for at least 6 months prior to study enrolment.

Exclusion Criteria:

* History or presence of cardiovascular, vascular, respiratory, renal, liver, musculoskeletal, endocrine, neuromuscular, metabolic, menstrual cycle and/or sleep related disease/disorder/dysfunction.
* Inability to perform exercise and pulmonary function testing.
* Taking doctor prescribed medication, other than oral contraceptives for women.
* Allergy to lidocaine or its 'caine' derivatives.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Exercise endurance time (EET) | Participants will be followed until all study visits are completed, an expected average of 2 weeks
  Exercise endurance time (EET) will be defined as the duration of loaded pedalling during constant work rate cycle exercise testing at 85% of each participants maximum incremental power output (in watts).
Esophageal temperature (in degrees Celsius) at isotime during exercise | Participants will be followed until all study visits are complete, an expected average of 2 weeks
  Esophageal temperature, recorded using an esophageal thermistor and estimating core body temperature, averaged over the last 30-secs of the highest equivalent exercise time (isotime) achieved by a given subject during exercise under the two treatment periods.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph.D., Principal Investigator — McGill University
Locations (1):
- McGill University, Dept. of Kinesiology & Physical Education, Clinical Exercise & Respiratory Physiology Laboratory, Montreal, Quebec, Canada

REFERENCES:
- See also: Clinical Exercise & Respiratory Physiology Laboratory (CERPL) of McGill University — http://www.mcgill.ca/cerpl